CLINICAL TRIAL: NCT00992420
Title: GIFT: Genotype Information and Functional Testing Study
Brief Title: Genotype Information and Functional Testing Study
Acronym: GIFT
Status: Completed | Type: Observational
Sponsor: Scripps Health (Other)
Collaborators: Bristol-Myers Squibb (Industry); Sanofi (Industry); Accumetrics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: P95082S
Record Dates: First submitted 2009-10-05; First posted 2009-10-09 (Estimated); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Coronary Artery Disease
Keywords: thienopyridine; platelets; CYP2C19; clopidogrel; platelet function tests; platelet; genes; cytochrome P450; single nucleotide polymorphisms; Platelet Aggregation Inhibitors
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- GRAVITAS Study Arm A: "Tailored" clopidogrel regimen - total first day dose 600-mg, then 150-mg every day for 6 months
- GRAVITAS Study Arm B: "Standard" clopidogrel regimen - a placebo loading dose (six placebo tablets) and then clopidogrel 75-mg and 1 placebo tablet every day for 6 months.
- GRAVITAS Study Arm C: Responders: A random sample of clopidogrel responders treated with a placebo loading dose (six placebo tablets) and then the standard clopidogrel regimen of 75-mg and 1 placebo tablet every day for 6 months.

SUMMARY:
This study is a sub-study of GRAVITAS (clinicaltrials.gov identifier NCT00645918). The purpose of this study is to assess which genes influence residual platelet reactivity on standard dose clopidogrel therapy, and also to determine whether certain genes influence the incremental change in platelet reactivity with high-dose clopidogrel maintenance dosing in patients who have high residual platelet reactivity on standard dosing.

DETAILED DESCRIPTION:
AS DESCRIBED BY THE PI: This study is a sub-study of GRAVITAS (clinicaltrials.gov identifier NCT00645918). The purpose of this study is to assess which genes influence residual platelet reactivity on standard dose clopidogrel therapy, and also to determine whether certain genes influence the incremental change in platelet reactivity with high-dose clopidogrel maintenance dosing in patients who have high residual platelet reactivity on standard dosing.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting inclusion criteria for GRAVITAS who undergo VerifyNow blood sampling for VerifyNow P2Y12 platelet function testing and IVRS entry for GRAVITAS randomization/selection determination

Exclusion Criteria:

* See GRAVITAS trial (ClinicalTrials.gov identifier: NCT00645918)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients meeting inclusion criteria for GRAVITAS who undergo VerifyNow blood sampling for VerifyNow P2Y12 platelet function testing and IVRS entry for GRAVITAS randomization/selection determination.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2009-10-01 (Actual); Primary Completion 2010-08-31 (Actual); Study Completion 2010-08-31 (Actual)

PRIMARY OUTCOMES:
residual platelet reactivity | 6 months
  Outcome 1 is residual platelet reactivity the measurement

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Price, MD, Principal Investigator — Scripps Clinic, La Jolla, CA
Locations (1):
- Scripps Genomic Medicine, La Jolla, California, United States

REFERENCES:
- [Derived] Price MJ, Murray SS, Angiolillo DJ, Lillie E, Smith EN, Tisch RL, Schork NJ, Teirstein PS, Topol EJ; GIFT Investigators. Influence of genetic polymorphisms on the effect of high- and standard-dose clopidogrel after percutaneous coronary intervention: the GIFT (Genotype Information and Functional Testing) study. J Am Coll Cardiol. 2012 May 29;59(22):1928-37. doi: 10.1016/j.jacc.2011.11.068. PMID 22624833